CLINICAL TRIAL: NCT05208892
Title: Dexmedetomidine Use in Suprazygomatic Maxillary Nerve Blocks for Pediatric Adenotonsillectomy Pain Control
Brief Title: Dexmedetomidine Use in SZMN Blocks for Pediatric T&A Pain Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stephanie Jiaying Pan, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 64309
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Opioid Use
Keywords: Suprazygomatic maxillary nerve block; Tonsillectomy and Adenoidectomy; Regional Anesthesia; Dexmedetomidine; Pediatric
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Patients in the two intervention groups will receive bilateral suprazygomatic maxillary nerve block such that 5 mL of local anesthetic is deposited on each side. Patients in the SZMN+Dexmedetomidine group will receive Dexmedetomidine in addition to the local anesthetic with placement of the suprazygomatic maxillary nerve block (0.25 mcg/kg on each side for a total dose of 5 mcg/kg, max 20 mcg total).
Who Masked: Participant, Care Provider
Masking Description: All three groups will receive a small circular band-aid on their temples (site of suprazygomatic maxillary nerve block placement).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SZMN Treatment Group (Experimental): Patients randomized into the SZMN treatment group will receive bilateral single injection SZMN blocks under general anesthesia in the operating room. The injection will occur through the pterygomaxillary fissure into the pterygomaxillary fossa. Patients will receive 5 ml of local anesthetic per side.
  Interventions: Procedure: SZMN block
- SZMN+Dexmedetomidine Treatment Group (Experimental): Patients randomized into the SZMN+Dexmedetomidine treatment group will receive bilateral single injection SZMN blocks under general anesthesia in the operating room. The injection will occur through the pterygomaxillary fissure into the pterygomaxillary fossa. Patients will receive 5 ml of local anesthetic along with 0.25 mcg/kg (max 10 mcg) Dexmedetomidine on each side (total of 0.5 mcg/kg, total max 20 mcg).
  Interventions: Procedure: SZMN block with Dexmedetomidine
- No Intervention: Control Group (No Intervention): Patients in this group will receive the standard of care for T&A procedures within the pediatric population.

INTERVENTIONS:
Procedure: SZMN block — Suprazygomatic Maxillary Nerve (SZMN) Blocks bilaterally
  Arms: SZMN Treatment Group
Procedure: SZMN block with Dexmedetomidine — Suprazygomatic Maxillary Nerve (SZMN) Blocks with local anesthetic and Dexmedetomidine bilaterally
  Arms: SZMN+Dexmedetomidine Treatment Group

SUMMARY:
The suprazygomatic maxillary nerve (SZMN) block is a well-established, safe and effective regional technique for pain management following cleft palate procedures. However, it has not been studied for patients undergoing tonsillectomy and adenoidectomy (T&A) procedures. The goal of this study is to determine whether the SZMN block can be utilized to improve pain control and decrease morbidity in pediatric patients undergoing T&A. An additional goal will be to determine whether the use of dexmedetomidine as a local anesthetic adjunct can prolong the analgesic effects of the SZMN block to cover the entire duration of pain experienced.

DETAILED DESCRIPTION:
Patients between 6 months and 18 years undergoing T&A surgical procedures will be reviewed for potential study enrollment. If participants agree to participate, they will be randomized into one of the three groups:

* the suprazygomatic maxillary nerve (SZMN) block treatment cohort
* the SZMN block with Dexmedetomidine treatment cohort
* the control cohort (standard of care).

After anesthesia induction, patients randomized into the SZMN-treatment group or SZMN+Dexmedetomidine treatment group will receive bilateral single injection SZMN blocks under general anesthesia in the operating room.

Participants enrolled into the control group will receive the standard of care with no changes to their anesthetic or surgical care. This group will not receive the SZMN block.

Postoperative pain scores and opioid consumption for all three groups will be collected in the PACU and for each postoperative day for a total of 14 postoperative days. We will also collect the following data: time to discharge readiness, postoperative nausea/vomiting, emergence delirium, oxygen desaturation and respiratory events, ability to tolerate oral intake, bleeding, hospital readmission, and adverse events related to the nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 months - 18 years
* Give consent/parental consent to participate in study
* Patients undergoing tonsillectomy and adenoidectomy

Exclusion Criteria:

* Participants who do not consent or have parental consent
* Patients who require urgent/emergent intervention
* Patients who undergo additional combined surgical procedures with separate incisions (in addition to the adenotonsillectomy)
* Patients with known difficult airway, clinical hemodynamic instability, coagulopathy, chronic pain history, chronic pain medication use, and unrepaired congenital heart disease
* Patients under age 6 months

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative Surgical Pain | Time Frame: 14 days after surgery
  Patients will rate their pain on a 0-10 scale
Postoperative Opioid Consumption | Time Frame: 14 days after surgery
  Amount of pain medications consumed by patients will be recorded

SECONDARY OUTCOMES:
Post-operative nausea, vomiting, delirium, ability to tolerate oral intake, bleeding, respiratory events, hospital readmission, time to discharge readiness | Time Frame: 14 days after surgery
  Adverse events following the procedure will be monitored and recorded
Complications from block | Time Frame: 14 days after surgery
  Nerve block complications will be monitored and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ban CH Tsui, MD, Study Director — Stanford University; Stephanie Pan, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Childrens Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grainger J, Saravanappa N. Local anaesthetic for post-tonsillectomy pain: a systematic review and meta-analysis. Clin Otolaryngol. 2008 Oct;33(5):411-9. doi: 10.1111/j.1749-4486.2008.01815.x. PMID 18983373
- [Background] Chiono J, Raux O, Bringuier S, Sola C, Bigorre M, Capdevila X, Dadure C. Bilateral suprazygomatic maxillary nerve block for cleft palate repair in children: a prospective, randomized, double-blind study versus placebo. Anesthesiology. 2014 Jun;120(6):1362-9. doi: 10.1097/ALN.0000000000000171. PMID 24525630